CLINICAL TRIAL: NCT05802901
Title: The Effect of Combining Spinal Manipulation and Dry Needling in Individuals With Non-specific Low Back
Brief Title: The Effect of Combining Spinal Manipulation and Dry Needling in Individuals With Low Back Pain
Acronym: SMTDNLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jedidiah Farley, Research Fellow, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 144339
Record Dates: First submitted 2023-03-07; First posted 2023-04-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Non-specific Low Back Pain
Keywords: Low back pain; Spinal manipulation; Dry needling; Diagnostic ultrasound; Oswestry disability index; Numeric pain rating scale
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal; Dry Needling

STUDY DESIGN:
Intervention Model Description: Three groups of participants receive one of three different interventions. One group receives spinal manipulation only, another group receives dry needling only, and the last group receives the combination of spinal manipulation and dry needling. Participants in each group receive their respective treatment in parallel with the other groups.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spinal manipulation (Active Comparator): Spinal manipulation of the lumbar spine only group.
  Interventions: Procedure: Spinal manipulation
- Dry needling (Active Comparator): Dry needling of the symptomatic side of the lumbar spine only group.
  Interventions: Procedure: Dry needling
- Spinal manipulation and dry needling (Active Comparator): Combination of spinal manipulation and dry needling of the lumbar spine group
  Interventions: Procedure: Spinal manipulation and dry needling

INTERVENTIONS:
Procedure: Spinal manipulation — Spinal manipulation of the lumbar spine only to be performed in the spinal manipulation arm/group.
  Arms: Spinal manipulation
Procedure: Dry needling — Dry needling of the lumbar erector spinae, multifidus, and gluteus medius on the symptomatic side performed in the dry needling arm/group.
  Arms: Dry needling
Procedure: Spinal manipulation and dry needling — The spinal manipulation and dry needling arm/group receive both spinal manipulation and dry needling as outlined in the other groups.
  Arms: Spinal manipulation and dry needling

SUMMARY:
The goal of this study is to enroll and randomize 99 participants with non-specific low back pain into a multimodal strategy of treatment consisting of a combination of dry needling (DN) and spinal manipulation therapy (SMT), DN only, and SMT only, followed by an at home exercise program. All groups will receive their respective treatment twice a week for 2 weeks followed by a 2-week home exercise program. Primary outcomes include clinical subjective (Oswestry Disability Index, numeric pain intensity rating) and mechanistic (lumbar multifidus, erector spinae, and gluteus medius muscle activation) measures assessed at baseline, 1, 2, and 4 weeks. Timepoints at 2-weeks and 4-weeks will be compared to baseline measures to determine effectiveness of the combination group against the other single treatment groups. Exercise compliance will be measured by participants self-reporting adherence to the program by selecting average number of days per week the exercises are completed.

ELIGIBILITY:
Inclusion Criteria:

* Presence of nonspecific low back pain defined as pain between the twelfth rib and buttocks with or without symptoms into one or both legs
* Current patient-reported pain rating score greater than 3 based on the numeric pain rating score 0-10 scale
* Oswestry Disability Index > 20%

Exclusion Criteria:

* Prior surgery to the lumbosacral spine
* Pregnancy
* Currently receiving mind-body or exercise treatment for low back pain with a healthcare provider (e.g., chiropractic, physical therapy, massage therapy, etc.)
* Signs of neurogenic low back pain arising from clinical examination (e.g., positive straight leg raise test, diminished muscle stretch reflex, etc.)
* Evidence of significant spinal pathology (e.g., spinal fracture, infection, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale at Baseline | Baseline
  Participants were asked to make separate ratings of current pain intensity and the best and worst intensity over the past 24 hours on a 0-10 scale ("0" no pain and "10" worst imaginable pain). The mean of the three ratings was used to represent pain intensity.
Low back pain Oswestry Disability Index Questionnaire at Baseline | Baseline
  The ODI score is derived from the Oswestry Disability Questionnaire, resulting in a score ranging from 0-100 with higher numbers indicating a greater level of disability.
Numeric pain rating scale at 1-week | 1-week
  Participants were asked to make separate ratings of current pain intensity and the best and worst intensity over the past 24 hours on a 0-10 scale ("0" no pain and "10" worst imaginable pain). The mean of the three ratings was used to represent pain intensity.
Low back pain Oswestry Disability Index Questionnaire at 1-week | 1-week
  The ODI score is derived from the Oswestry Disability Questionnaire, resulting in a score ranging from 0-100 with higher numbers indicating a greater level of disability.
Numeric pain rating scale at 2-weeks | 2-weeks
  Participants were asked to make separate ratings of current pain intensity and the best and worst intensity over the past 24 hours on a 0-10 scale ("0" no pain and "10" worst imaginable pain). The mean of the three ratings was used to represent pain intensity.
Low back pain Oswestry Disability Index Questionnaire at 2-weeks | 2-weeks
  The ODI score is derived from the Oswestry Disability Questionnaire, resulting in a score ranging from 0-100 with higher numbers indicating a greater level of disability.
Numeric pain rating scale at 4-weeks | 4-weeks
  Participants were asked to make separate ratings of current pain intensity and the best and worst intensity over the past 24 hours on a 0-10 scale ("0" no pain and "10" worst imaginable pain). The mean of the three ratings was used to represent pain intensity.
Low back pain Oswestry Disability Index Questionnaire at 4-weeks | 4-weeks
  The ODI score is derived from the Oswestry Disability Questionnaire, resulting in a score ranging from 0-100 with higher numbers indicating a greater level of disability.

SECONDARY OUTCOMES:
Lumbar multifidus muscle change in thickness at Baseline | Baseline
  Muscle activation measured by changes in contraction thickness at rest and sub-maximal isometric contraction utilizing diagnostic ultrasound.
Erector spinae muscle change in thickness at Baseline | Baseline
  Muscle activation measured by changes in contraction thickness at rest and sub-maximal isometric contraction utilizing diagnostic ultrasound.
Gluteus medius muscle change in thickness at Baseline | Baseline
  Muscle activation measured by changes in contraction thickness at rest and sub-maximal isometric contraction utilizing diagnostic ultrasound.
Lumbar multifidus muscle change in thickness at 2-weeks | 2-weeks
  Muscle activation measured by changes in contraction thickness at rest and sub-maximal isometric contraction utilizing diagnostic ultrasound.
Erector spinae muscle change in thickness at 2-weeks | 2-weeks
  Muscle activation measured by changes in contraction thickness at rest and sub-maximal isometric contraction utilizing diagnostic ultrasound.
Gluteus medius muscle change in thickness at 2-weeks | 2-weeks
  Muscle activation measured by changes in contraction thickness at rest and sub-maximal isometric contraction utilizing diagnostic ultrasound.
Lumbar multifidus muscle change in thickness at 4-weeks | 4-weeks
  Muscle activation measured by changes in contraction thickness at rest and sub-maximal isometric contraction utilizing diagnostic ultrasound.
Erector spinae muscle change in thickness at 4-weeks | 4-weeks
  Muscle activation measured by changes in contraction thickness at rest and sub-maximal isometric contraction utilizing diagnostic ultrasound.
Gluteus medius muscle change in thickness at 4-weeks | 4-weeks
  Muscle activation measured by changes in contraction thickness at rest and sub-maximal isometric contraction utilizing diagnostic ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Jedidiah Farley, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farley J, Taylor-Swanson L, Koppenhaver S, Thackeray A, Magel J, Fritz JM. The Effect of Combining Spinal Manipulation and Dry Needling in Individuals With Nonspecific Low Back Pain. J Pain. 2024 Aug;25(8):104506. doi: 10.1016/j.jpain.2024.03.002. Epub 2024 Mar 12. PMID 38484853

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT05802901/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT05802901/ICF_001.pdf